CLINICAL TRIAL: NCT02233673
Title: Incentives Targeting Gestational Weight Gain in Overweight/Obese Low Income Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Julie Phillips, Project Director, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-276
Record Dates: First submitted 2014-09-03; First posted 2014-09-08 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Overweight; Obesity; Pregnancy
Keywords: Obesity; Pregnancy
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral, incentives (Experimental): Participants receive behavioral intervention and financial incentives for meeting gestational weight gain goals
  Interventions: Behavioral: Financial incentives
- Standard care (No Intervention): Participants receive standard obstetrical care from their provider

INTERVENTIONS:
Behavioral: Financial incentives — Participants receive a behavioral intervention and financial incentives for meeting gestational weight gain goals.
  Arms: Behavioral, incentives

SUMMARY:
Excessive weight gain during pregnancy, particularly in overweight and obese women, predisposes to adverse perinatal outcomes and has long term effects on maternal and neonatal health. With an inverse relationship between socioeconomic status and obesity, significant health disparities exist between obese and normal weight women. The Institute of Medicine (IOM) recently revised its gestational weight gain recommendations, targeted to pregravid body mass index (BMI), to minimize pregnancy complications. However, these recommendations are based on cross sectional observational studies and neither the ideal method to achieve weight gain goals nor whether perinatal outcome is optimized with active management of weight gain is known. The investigators propose to investigate a behavioral incentive-based intervention to improve compliance with IOM weight gain recommendations during pregnancy in low-income overweight and obese women. The investigators will evaluate if 1) gestational weight gain can be reliably targeted to the IOM recommendations and 2) active weight gain management during pregnancy improves perinatal outcomes. Two study groups will be compared in a prospective randomized trial; 1) those receiving standard obstetrical care and 2) those receiving behavioral weight management counseling plus financial incentives for achieving weight gain goals. The main outcome measure will be the percentage of women gaining within the IOM recommendations based on prepregnancy BMI. Secondary outcomes evaluated will include fetal growth and body composition changes, birth weight and the rate of cesarean delivery. The investigators hypothesize that 1) the behavioral intervention with incentives will result in greater compliance to IOM guidelines for gestational weight gain than standard care and 2) targeting weight gain to the IOM guidelines will lead to a reduction in the rates of fetal macrosomia and cesarean delivery. Finally, cost effectiveness of treatment conditions will be examined. This intervention, if efficacious and cost-effective, has the potential to improve compliance with gestational weight gain guidelines, optimize perinatal outcomes, and reduce health disparities.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years of age and ≤ 45 years of age

-≤16 weeks gestation

* BMI ≥25
* Ultrasound documented viable singleton intrauterine pregnancy
* English speaking
* Planning to deliver at Fletcher Allen Health Care
* Willing to be randomized to one of the study groups
* Written informed consent

Exclusion Criteria:

* Major fetal congenital or chromosomal anomaly
* Women with a restricted diet (i.e., celiac disease, prior bariatric surgery, Phenylketonuria, or other metabolic disorder)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2014-03; Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain within the Institute of Medicine guidelines | At time of delivery
  Total gestational weight gain at time of last prenatal visit. For participants in the intervention arm, gestational weight gain at 2 week intervals will also be assessed.

SECONDARY OUTCOMES:
Cesarean delivery rate | Time of delivery
  Cesarean delivery rate (as a percent of total deliveries) will be assessed
Fetal macrosomia | At delivery
  Fetal weight at delivery will be recorded. Percent fetal macrosomia (birthweight >4000g) will be assessed.

OTHER OUTCOMES:
Cost of intervention | Intake to 6 weeks postpartum
  Costs to the patient attending the intervention (transportation, childcare, missed wages) will be calculated against cost differences in outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Derived] Phillips JK, Skelly JM, Roberts LM, Bernstein IM, Higgins ST. Combined financial incentives and behavioral weight management to enhance adherence with gestational weight gain guidelines: a randomized controlled trial. Am J Obstet Gynecol MFM. 2019 Mar;1(1):42-49. doi: 10.1016/j.ajogmf.2019.02.002. Epub 2019 Mar 5. PMID 33319756